CLINICAL TRIAL: NCT04101955
Title: Ultrasound Guided - Incisionless Thread Carpal Tunnel Release Versus Standard Mini-Open Carpal Tunnel Release for the Treatment of Carpal Tunnel Syndrome: A Randomized Trial
Brief Title: Ultrasound Guided - Incisionless Threaded Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander Y. Shin, M.D., M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-010569
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incisionless Threaded Carpal Tunnel (Other)
  Interventions: Procedure: Incisionless Threaded Carpal Tunnel; Procedure: Standard Mini-Open Carpal Tunnel
- Standard Mini-Open Carpal Tunnel (Other)
  Interventions: Procedure: Incisionless Threaded Carpal Tunnel; Procedure: Standard Mini-Open Carpal Tunnel

INTERVENTIONS:
Procedure: Incisionless Threaded Carpal Tunnel — ultra-minimally invasive thread carpal tunnel release
Procedure: Standard Mini-Open Carpal Tunnel — open surgical carpal tunnel release

SUMMARY:
The overarching long-term goal is to develop a CTS Treatment Center within the Hand Clinic that offers a variety of established and emerging treatment options in a multidisciplinary program. The ultra-minimally invasive carpal tunnel release would be one component of the program. Furthering the knowledge with regard to ultra-minimally invasive carpal tunnel release outcomes would facilitate the Hand Clinics ability to offer this procedure as a component of individualized care in the CTS Treatment Center to facilitate delivery of the appropriate level of care to the right patient.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CTS with symptoms including pain, paresthesia's, and weakness of the hand in the median nerve distribution for minimum of 3 months
* Age 18-65 years old
* Persistence of symptoms after 6 weeks of conservative treatment such as splinting, activity modification, and/or injection therapy.
* Electromyographic evidence of mild, moderate, moderately severe, or severe median nerve neuropathy at the wrist
* Ability to complete all follow up appointments

Exclusion Criteria:

* Previous CTS surgical release on affected side
* Diabetes mellitus
* Hypothyroidism
* Hand arthritis (rheumatologic or osteoarthritis)
* Pregnancy
* Electromyographic evidence of any condition other than CTS affecting the hand
* Workman's compensation
* Participants not willing to make follow-up visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) functional score | Time Frame: Change from Baseline to 12 months
  Measured on a symptom severity scale from 1 to 5, where 1 is normal and 5 is very serious/continued/difficult
Visual analog pain scale | Time Frame: Change from Baseline to 12 months
  Pain that participant is currently experiencing the in the hand or risk(0-100)
Strength testing of grip | Time Frame: Change from Baseline to 12 months
  Use dynameters
Disability of the Arm Shoulder Hand DASH | Time Frame: Change from Baseline to 12 months
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The main purpose of this study was to assess the longitudinal construct validity of the DASH among patients undergoing surgery. The second purpose was to quantify self-rated treatment effectiveness after surgery.
Strength testing of pinch | Time Frame: Change from Baseline to 12 months
  Use pinch meters

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papanicolaou GD, McCabe SJ, Firrell J. The prevalence and characteristics of nerve compression symptoms in the general population. J Hand Surg Am. 2001 May;26(3):460-6. doi: 10.1053/jhsu.2001.24972. PMID 11418908
- [Background] Harry S, Tanya R. Carpal tunnel claims rank second among major lost time diagnosis. NCCI Research Brief 2005 Apr; Vol.3
- [Background] Fajardo M, Kim SH, Szabo RM. Incidence of carpal tunnel release: trends and implications within the United States ambulatory care setting. J Hand Surg Am. 2012 Aug;37(8):1599-605. doi: 10.1016/j.jhsa.2012.04.035. Epub 2012 Jun 23. PMID 22727925
- [Background] Huisstede BM, Hoogvliet P, Randsdorp MS, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part I: effectiveness of nonsurgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):981-1004. doi: 10.1016/j.apmr.2010.03.022. PMID 20599038
- [Background] Huisstede BM, Randsdorp MS, Coert JH, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part II: effectiveness of surgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):1005-24. doi: 10.1016/j.apmr.2010.03.023. PMID 20599039
- [Background] Guo D, Guo D, Guo J, Malone DG, Wei N, McCool LC. A Cadaveric Study for the Improvement of Thread Carpal Tunnel Release. J Hand Surg Am. 2016 Oct;41(10):e351-e357. doi: 10.1016/j.jhsa.2016.07.098. Epub 2016 Aug 20. PMID 27554942
- [Background] Guo D, Guo D, Guo J, Schmidt SC, Lytie RM. A Clinical Study of the Modified Thread Carpal Tunnel Release. Hand (N Y). 2017 Sep;12(5):453-460. doi: 10.1177/1558944716668831. Epub 2016 Sep 12. PMID 28832215
- [Background] Guo D, Tang Y, Ji Y, Sun T, Guo J, Guo D. A non-scalpel technique for minimally invasive surgery: percutaneously looped thread transection of the transverse carpal ligament. Hand (N Y). 2015 Mar;10(1):40-8. doi: 10.1007/s11552-014-9656-4. PMID 25767420
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Greenslade JR, Mehta RL, Belward P, Warwick DJ. Dash and Boston questionnaire assessment of carpal tunnel syndrome outcome: what is the responsiveness of an outcome questionnaire? J Hand Surg Br. 2004 Apr;29(2):159-64. doi: 10.1016/j.jhsb.2003.10.010. PMID 15010164
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials